CLINICAL TRIAL: NCT03915717
Title: Observational Study of Outcomes After EchoMark and EchoSure-based Free Flap Monitoring
Status: Terminated | Type: Observational
Why Stopped: Slow Enrollment
Sponsor: Sonavex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-01
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Free Flap Transfer; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EchoMark — EchoMark is implanted during surgery to mark the at-risk blood vessels to enable EchoSure ultrasound-based monitoring
Device: EchoSure — EchoSure ultrasound scans are performed to monitor the free flap

SUMMARY:
The purpose of this study is to evaluate the performance of the EchoMark and EchoSure as an ultrasound-based method of monitoring the viability of free flaps and patency of at-risk vessels.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients presenting for microvascular tissue transfer procedures where the surgeon has selected EchoMark and EchoSure as the optimal method of vascular monitoring based on clinical assessment and plan
* Patient is able to sign informed consent and able to participate in all testing associated with this clinical investigation
* Women of childbearing potential have a negative pregnancy test

Exclusion Criteria:

* Age <18 years old
* Patient unable to sign informed consent
* Patient participating in another investigational device or pharmacological study
* Prisoner or patient from vulnerable populations as defined in 45 CFR 46.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing free flap surgery
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EchoMark / EchoSure: Patients undergoing free flap surgery and have an EchoMark soft tissue marking device placed and monitored with the EchoSure.
Period: Overall Study
Arm/Group | EchoMark / EchoSure
Started | 14
Completed | 8
Not Completed | 6
Not completed — EchoMark Not Implanted | 6

BASELINE CHARACTERISTICS:
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: Years] | 64 [55 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Surgeon Evaluation of Improved Monitoring Ability Via Questionnaire With Likert Scale
Description: Surgeon evaluation of improved monitoring ability via questionnaire with likert scale
Time Frame: Through study completion
Population: Surgeon Evaluation Questionnaire was not completed, Data was not collected.
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 0

2. Primary Outcome: Surgeon Evaluation of Satisfaction
Description: Surgeon evaluation of satisfaction via questionnaire with likert scale
Time Frame: Through study completion, an average of 1 year
Population: Surgeon Satisfaction Survey was not completed. Data not collected.
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 0

3. Secondary Outcome: Flap Failure Rate
Description: Percentage of flaps that fail
Time Frame: Through patient stay, up to 5 days post-op
Measure: Number; unit: Flaps that Failed
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 8
Flaps that Failed | 0

4. Secondary Outcome: Flap Takeback Rate
Description: Percentage of flaps that require return to the OR after the baseline procedure through 5 days post-op.
Time Frame: Through patient stay, up to 5 days post-op
Measure: Number; unit: Flaps that Required Return to the OR
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 8
Flaps that Required Return to the OR | 0

5. Secondary Outcome: Flap Salvage Rate
Description: Percentage of flaps that require salvage after the baseline procedure
Time Frame: Through patient stay, up to 5 days post-op
Measure: Number; unit: Number of Flaps that Require Salvage
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 8
Number of Flaps that Require Salvage | 0

6. Secondary Outcome: Total Cost of Hospitalization
Time Frame: Through patient stay, up to 5 days post-op
Population: Data was not collected on hospitalization costs.
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 0

7. Secondary Outcome: Time From OR Departure to Return to OR
Description: Number of hours from when the subject's baseline procedure ends until a secondary trip to the OR if required.
Time Frame: Through patient stay, up to 5 days post-op
Measure: Mean (Full Range); unit: Hours
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 8
Hours | NA [NA to NA] — Time to return to OR cannot be calculated due to insufficient number of participants with events

8. Secondary Outcome: Nurse Evaluation of Improved Monitoring Via Questionnaire With Likert Scale
Time Frame: Through study completion, an average of 1 year
Population: The Nurse Questionnaire was not completed. Data was not collected.
Arm/Group | EchoMark / EchoSure
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected from the baseline procedure until discharge, an average of 72 hours.
Arm/Group | EchoMark / EchoSure
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT03915717/Prot_SAP_000.pdf